CLINICAL TRIAL: NCT01342705
Title: Influence of Iron Depletion by Phlebotomy on the Risk of Hepatocellular Carcinoma Occurrence in Patients With Compensated Alcoholic Cirrhosis. Prospective, Multicentre, Randomized Trial
Brief Title: Phlebotomy and Risk of Hepatocellular Carcinoma in Patients With Compensated Alcoholic Cirrhosis
Acronym: CIRROX
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: delayed recruitment as compared to that expected
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P091107
Record Dates: First submitted 2011-04-14; First posted 2011-04-27 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2012-11

CONDITIONS: Alcoholic Cirrhosis; Iron Overload
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Iron Overload | interventions — Phlebotomy; Bloodletting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- phlebotomy (Experimental)
  Interventions: Procedure: phlebotomy
- control (No Intervention)

INTERVENTIONS:
Procedure: phlebotomy — Procedure: Phlebotomy of 4 ml / kg to obtain (1 phlebotomy every 14 days) and maintain (1 phlebotomy every 3 months) a serum ferritin below 50 µg / l.
  Other Names: Bloodletting; Iron depletion
  Arms: phlebotomy

SUMMARY:
The main objective of the study is to assess in patients with compensated alcoholic cirrhosis and hepatic iron overload (HIO), as assessed by MRI, the effect of phlebotomy in order to lower and maintain serum ferritin below 50 µg / l on the risk of hepatocellular carcinoma (HCC) occurrence. The effect of bloodletting will be jointly evaluated on 1) episodes of hepatic decompensation, 2) non HCC liver-related mortality 3) changes in HIO during follow-up.

DETAILED DESCRIPTION:
Purpose

The role of iron in liver carcinogenesis is supported by human, animal and cellular models through direct and indirect mechanisms. The accumulation of iron promotes liver cell proliferation and is responsible for direct structural damage or mutations of DNA caused by free iron itself or reactive oxygen species generated by its accumulation in the liver.

The influence of hepatic iron overload (HIO) on the risk of hepatocellular carcinoma (HCC) is well established in patients with genetic hemochromatosis or HCC developed on non-cirrhotic liver. However, the influence of HIO on the risk of occurrence of HCC in other chronic liver disease (including alcoholic and viral C) has been controversial. Recently, a prospective study including a large population of patients with cirrhosis (n = 301) classified according to the aetiology of liver disease (alcohol, n = 162 or hepatitis C virus (HCV)infection, n = 139) has shown the association between HIO and the occurrence of HCC in patients with alcoholic cirrhosis. Thus, the assessment of liver iron in routine clinical practice could allow the identification of patients at higher risk of developing HCC and in whom preventive measures such as iron depletion by phlebotomy could be undertaken. Based on the model of genetic hemochromatosis in which its effectiveness on survival improvement and even regression of hepatic injury has been shown, its effectiveness on the prognosis and prevention of HCC occurrence in patients with alcoholic cirrhosis must now be studied in prospective multicentre randomized trials.

The main objective of the study is to assess in patients with compensated alcoholic cirrhosis and HIO, as assessed by MRI, the effect of phlebotomy in order to lower and maintain serum ferritin below 50 µg / l on the risk of HCC occurrence. The effect of bloodletting will be jointly evaluated on 1) episodes of hepatic decompensation, 2) non HCC liver-related mortality 3) changes in HIO during follow-up.

Study Type: Interventional Study Design: Allocation: Randomized Endpoint Classification: Efficacy Study Intervention Model: Parallel Assignment Masking: Open Label Primary Purpose: Prevention

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Biopsy-proven alcoholic cirrhosis
* No previous HCC (treated or not)
* Excessive alcohol consumption, defined by more than 21 glasses weekly in women and more than 28 glasses weekly in men for at least 10 years, and considered as the main cause for liver cirrhosis
* Signed written informed consent
* Hepatic iron overload assessed by MRI (Iron hepatic concentration ≥ 80 μmol/g)

Exclusion Criteria:

* Subjects deprived of their liberty by judicial or administrative decision
* Pregnant women
* Serious associated short-term life threatening disease (except HIV viral co-infection, or the liver disease itself)
* Impossibility of monitoring, whatever the reason.
* Contraindication of phlebotomy
* Haemoglobin <13.5 g/dL for men and <12.5g/dL for women (threshold established by the French Blood Agency)

  * Congestive heart failure or coronary heart disease
  * Hepatic failure (TP<60%), renal failure (GFR <50 ml/min) or respiratory insufficiency (chronic dyspnea)
  * Poor venous system
* Complication of cirrhosis at time of inclusion (defined as bleeding related to portal hypertension, encephalopathy or ascites)
* Presence of hepatitis B or hepatitis C co-infection
* Presence of liver focal lesion suggestive of HCC
* Child-Pugh score greater than or equal to 7 (Class B or C) at time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of HepatoCellular Carcinoma during follow-up | 3 years
  the cumulative incidence of HCC will be estimated considering death prior to the event of interest as competing risk outcomes

SECONDARY OUTCOMES:
Number of hepatic decompensation episodes in study participants | 3 years
Cumulative incidence of death non related to hepatoCellular Carcinoma | 3 years
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierre NAHON, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (14):
- France (14):
  - Amiens University Hospital :, Amiens
  - Avicenne, Bobigny
  - Jean Verdier, Bondy
  - CHU Bordeaux univerity hospital 1, Bordeaux
  - CHU Bordeaux University hospital 2, Bordeaux
  - CHU, Caen
  - Antoine Béclère, Clamart
  - CHU, Grenoble
  - CHU, Lille
  - CHU, Montpellier
  - CHU, Nancy
  - CHU, Nice
  - CHU, Rennes
  - CHU, Rouen